CLINICAL TRIAL: NCT05294120
Title: A Phase II Trial of Reflectance ConfocaL Microscopy And Optical Coherence Tomography Guided RadIation TherapY: CLARITY
Brief Title: A Study on Radiation Therapy Guided by the Reflectance Confocal Microscopy (RCM)/Optical Coherence Tomography (OCT) Device in People With Basal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Physical Sciences Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-553
Record Dates: First submitted 2022-03-15; First posted 2022-03-24 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Basal Cell Carcinoma
Keywords: Radiation Therapy; Reflectance Confocal Microscopy (RCM)/Optical Coherence Tomography (OCT); 20-553
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, single-center, phase II, single-arm clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Reflectance ConfocaL Microscopy And Optical Coherence Tomography Guided RadIation Therapy (Experimental): If eligible, patients will undergo pretreatment RCM/OCT imaging, followed by RT.
  Six weeks after the completion of RT, patients will undergo post-treatment assessment with RCM/OCT and biopsy. If residual carcinoma is detected on the biopsy, surgical excision of the BCC will be performed. If no residual carcinoma is detected on the biopsy, the patient will be monitored for clinical evidence of recurrence for up to 3 years.
  Interventions: Device: Reflectance ConfocaL Microscopy And Optical Coherence Tomography Guided; Radiation: Radiation Therapy

INTERVENTIONS:
Device: Reflectance ConfocaL Microscopy And Optical Coherence Tomography Guided — Patients will undergo RCM/OCT with an imaging specialist in the Dermatology Service.
  This is not expected to take longer than 30 minutes. Prior to imaging, a digital photograph will be taken of the biopsy proven BCC.
Radiation: Radiation Therapy — After the completion of skin imaging, patients will undergo simulation and tumor radiotherapy. An equivalent total dose in 2 Gy fractions (EQD2) of 45-46 Gy will be delivered for treatment.

SUMMARY:
The purpose of this study is to find out if radiation therapy (RT) guided by the new reflectance confocal microscopy (RCM)/optical coherence tomography (OCT) device is an effective treatment for basal cell carcinoma (BCC). The researchers will also look at the side effects from RT guided by the RCM/OCT device. In addition, will determine the quality of life before and after treatment by having the participant fill out questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven basal cell carcinoma

  °Up to 3 tumors per patient can be treated per protocol synchronously or metachronously
* Clinical stage T1 or T2 by Union International to Control Cancer 8th edition system

  * ≤40 mm in maximum dimension
  * no deep invasion (beyond subcutaneous fat or >6 mm from granular later of dermis to deepest point of carcinoma)
  * no perineural invasion of nerves ≥0.1 mm diameter or deeper than dermis
  * no intraneural invasion
  * no bone erosion, invasion or foraminal transgression NOTE: For the purposes of protocol inclusion, if any of the features mentioned above is not included in the pathology report they will considered absent.
* ≥18 years old
* Amenable to RCM/OCT and radiation therapy in opinion of investigator

  * Some anatomic locations may preclude imaging by RCM/OCT may not be amenable to RCM/OCT imaging
  * Some medical comorbidities may preclude the delivery of radiation therapy (conditions rendering patients hypersensitive to ionizing radiation, or unable to undergo treatment)
* Able and willing to complete the Skindex 16 and Skin Cancer Index (must be able to understand English or Spanish)

Exclusion Criteria:

* Medical contraindication to radiation therapy in the opinion of the investigator
* Prior cancer radiotherapy which precludes the ability to safely deliver radiation therapy in the opinion of the investigator
* High likelihood of protocol non-compliance in the opinion of the investigator °Patients who demonstrate unwillingness to undergo protocol-defined treatment or follow-up procedures will be ineligible to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
histologic tumor response rate | 6 weeks
  The presence of residual carcinoma on a biopsy or surgical excision specimen will be primary determinant for the primary endpoint outcome.

SECONDARY OUTCOMES:
frequency and severity of adverse events | up to 12 weeks
  by the Common Terminology and Criteria for Adverse Events, version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

DOCUMENTS (1):
  • Informed Consent Form (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/20/NCT05294120/ICF_000.pdf